CLINICAL TRIAL: NCT03072693
Title: Daily Ambulatory Remote Monitoring System Vs Conventional Therapy For The Post-Dischage Management Of Acute Decompensated Heart Failure
Brief Title: Daily Ambulatory Remote Monitoring System For Post-Dischage Management Of ADHF
Acronym: DAVID-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other); Novartis Pharmaceuticals (Industry); Biofourmis Singapore Pte Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Chung-Wah David SIU, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARDIAC_HF_1
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Remote monitoring device given to subjects for daily monitoring to vital signs, activities and discomfort. Medication to be adjusted by investigators according to the recorded parameters and patients' condition.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Home-based remote heart failure management
  Interventions: Procedure: Home-based remote heart failure management
- Group 2 (Placebo Comparator): Home-based physiological parameter recording only
  Interventions: Procedure: Home-based physiological parameter recording only

INTERVENTIONS:
Procedure: Home-based remote heart failure management — For patients randomized to Group 1, the home-based remote heart failure management system will be connected via the internet for active intervention. In Group 2 patients, the system will not be activated although all data will continue to be stored and reviewed at clinic visits. For patients in Group 1, clinically-assigned targets and alert thresholds of individual physiological parameters including blood pressure, pulse rate, and body weight will be decided before discharge and at entry into the three management modes. Site investigators will review individual patient physiological parameters upon clinic visits, and treatment can be initiated through instant communication (electronic communication and/or phone).
  Arms: Group 1
Procedure: Home-based physiological parameter recording only — For patients randomized to Group 2, the home-based remote heart failure management system will continuously record and store patients information to be reviewed at clinic visits but not connected to internet. Site investigators will review individual patient physiological parameters upon clinic visits, and no treatment will be initiated through instant communication.
  Arms: Group 2

SUMMARY:
Background: Despite the advances in pharmacological management of heart failure (HF), the associated mortality and re-hospitalization for HF remain poor. This is at least partly due to suboptimal early discharge care, delayed detection of HF complications, and underutilization and under-dosing of evidence-based HF medications. Mobile technology has revolutionized inter-personal communication allowing instantaneous, multi-directional, and massive data transfer. Nonetheless the potential of these enhanced communications have not been fully explored in the management of patients with HF.

Objective: To explore the potential of state-of-the-art mobile technology for home-based remote HF management in order to reduce HF mortality and HF re-hospitalization.

Study Design: This will be a multicenter, randomized controlled clinical trial in patients with HF and reduced left ventricular ejection fraction (LVEF) who are discharged from hospital following an episode of acutely decompensated HF. The clinical effectiveness of a physician-directed patient self-management strategy based on remotely collected physiological data obtained from home-based and wearable devices will be compared with two control groups who will receive the home-based remote HF management system without activation or routine therapy. In the interventional arm, there will be three modes of home-based HF management: (1) Early discharge mode to optimize volume status; (2) Drug escalation mode to ensure the utilization of evidence-based medications at the maximum tolerated dose; and (3) Maintenance mode to ensure medication compliance and early detection of complications such as acutely decompensated HF and atrial fibrillation. The trial will enroll up to 876 patients with LVEF <40% who are discharged from hospital after an episode of acutely decompensated HF. Randomization to the intervention group or control groups will be in a 1:1:1 ratio with follow-up for 1 year. The primary outcome will be a composite of cardiovascular death and HF hospitalization within 1 year.

Summary: DAVID-HF will provide essential information about the role of home-based, remote heart failure monitoring that will incorporate instantaneous physician-directed patient-self management in the long-term management of HF patients.

DETAILED DESCRIPTION:
METHODS Study Design DAVID-HF is a prospective, multi-center, randomized controlled, open-labeled study. The study is registered with the ClinicalTrials.gov. Patients with acutely decompensated HF and reduced LVEF on discharge from hospital will be randomized in a 1:1:1 ratio to home-based remote HF management system with active physician-directed management or home-based remote HF management without activation or optimal medical management (routine care). (Figure 1) The investigation conforms with the principles outlined in the Declaration of Helsinki. The study protocol has been approved by the Institutional Review Board of The University of Hong Kong, and Hong Kong West Cluster, Hospital Authority, Hong Kong. Approval at other participating sites will be subsequently obtained.

Patients The patient eligibility criteria are summarized in Table 1. Briefly, adult patients discharged from hospital following an episode of acutely decompensated HF that required intravenous diuretic therapy within 14 days and with LVEF <40% will be recruited. The diagnosis of ADHF will be based on (1) the presence of symptoms and signs of heart failure as defined according to the Framingham Heart Failure Score (≥2) at the time of admission, (Table 2)(17) (2) radiographic evidence of pulmonary congestion on chest radiography, and (3) elevated serum concentration of brain-type natriuretic peptide (BNP) >100 pg/mL. Patients will be excluded if they have a history of acute coronary syndrome within the last four weeks, complex congenital heart disease, or significant valvular stenosis, are unable to operate simple electronic devices, are unable or refuse to provide informed consent, or if a mobile network service is unavailable in the place of residence.

Home-based Remote Heart Failure Management System The home-based remote heart failure management system has been designed and manufactured by Heartisans limited (Hong Kong SAR, China) in collaboration with Prof. Chung-Wah SIU from The University of Hong Kong. The system is able to remotely monitor a patient's physiological parameters that will be communicated wirelessly via a smartphone-based device to the heart failure team. (Figure 2) The system comprises a wearable heart failure monitor, a Blue-tooth blood pressure measuring device, and a Blue-tooth bath scale. The wearable heart failure monitor is capable of (1) photoplethysemograph (PPG)-based continuous pulse rate monitoring, (2) electrocardiogram (ECG) acquisition, (3) bio-impedance measurement, and has (4) an activity sensor in a wristband, and (5) a global positioning system (GPS)-based 6-minute walking distance test with a smartphone. The PPG-based pulse rate monitor will continuously acquire beat-to-beat RR Intervals with an intelligent motion artifact removal algorithm. The daily activity as detected by the motion sensor will continuously monitor patient activity. Patients will be instructed to record a 30-second single lead ECG and to perform one bio-impedance measurement every morning as well as to perform a 6-minute walking distance test every week. The wearable monitors will be worn for 16-18 hours during waking hours and be recharged while sleeping. In addition, patients will be instructed to measure their blood pressure in the morning and evening and body weight in the evening, every day. All remotely obtained physiological data will be transferred in real time through a specially-designed application on the smartphone to the doctor console. (Figure 3 and Table 3) All patients will be followed up for 1 year. (Table 4)

Intervention procedure After randomization, patients in Group 1 and Group 2 will be provided with a home-based remote heart failure management system, and will be instructed to perform daily routine measurements. (Table 3) For patients randomized to Group 1, the home-based remote heart failure management system will be connected via the internet for active intervention. In Group 2 patients, the system will not be activated although all data will continue to be stored and reviewed at clinic visits. For patients in Group 1, clinically-assigned targets and alert thresholds of individual physiological parameters including blood pressure, pulse rate, and body weight will be decided before discharge and at entry into the three management modes (see below). Site investigators will review individual patient physiological parameters upon clinic visits, and treatment can be initiated through instant communication (electronic communication and/or phone). Patients in Group 3 will receive routine care.

Early discharge mode The objective of early discharge is to optimize volume status, primarily using an oral diuretic. This will be accomplished by daily measurement of body weight, blood pressure, heart rate, and symptom score. Dosage of diuretic will be titrated as appropriate. (Appendix A)

Drug escalation mode The objective of drug escalation is to ensure the utilization of evidence-based medications at the maximally tolerated dose. These include angiotensin-converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), beta-adrenergic block (BB), mineralocorticoid antagonist (MRA), ivabradine, and sacubitril/valsartan. The aim is to maximize the dosage of one evidence-based anti-heart failure medication per week in a sequence according to European Society of Cardiology guidelines for the diagnosis and treatment of acute and chronic heart failure, i.e., first line: ACEI/ARB, MRA, and BB; and second line: ivabradine and sacubitril/valsartan.(18) The dosage of medications will be stepwise increased to the maximally tolerated dose according to patient status. (Appendix B) The duration of drug escalation will range from 2 to 16 weeks. Blood pressure, heart rate, body weight, subjective symptom score, daily activity, and 6-minute walking distance will be monitored.

Maintenance mode The objective of maintenance mode is to ensure medication compliance and early detection of complications such as acutely decompensated HF and atrial fibrillation. This will be accompanied by daily measurement of blood pressure, heart rate, body weight, subjective symptoms, daily activity, and single-lead ECG. (Appendix C)

Study measures The primary outcome measure will be a composite of re-hospitalization for acute decompensated HF and/or mortality within 1 year. The secondary outcomes will include 1-year mortality and 1-year re-hospitalization for acute decompensated HF rate, New York Heart Association functional class, average visual analogue symptom score, 6-minute walking distance, daily activity, utilization of evidence-based anti-HF medication, and quality of life measured with the Minnesota Living with Heart Failure questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Recently discharged from hospital for acutely decompensated HF (within 2 weeks) requiring intravenous diuretic therapy.
* Left ventricular ejection fraction <40%
* Voluntarily agrees to participate by providing written informed consent

Exclusion Criteria:

* Acute coronary syndrome within 4 weeks
* Complex congenital heart disease
* Significant valvular stenosis
* Left ventricular assist device
* Planned cardiac intervention including revascularization, cardiac resynchronization, and valvular surgery
* Listed for heart transplant
* Renal impairment with serum creatinine ≥250 μmol/L or on renal replacement therapy
* Inability or refusal to provide inform consent
* Lack of skills in operating simple electronic devices
* Unavailability of a mobile network service in the place of residence

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Composite Primary Endpoints | 12 months
  composite of re-hospitalization for acute decompensated HF and/or mortality

SECONDARY OUTCOMES:
1-year mortality | 12 months
  1-year mortality
1-year heart failure rehospitalization | 12 months
  1-year heart failure rehospitalization
Visual analog symptom score | Continuously for 12 months
  Visual analog symptom score for heart failure
6-minute walking distance | intermittently for 12 months
  6-minute walking distance
Utilization of evidence-based anti-heart failure medications | 12 months
  The number and percentage dosage of anti-heart failure medications
Quality of life | 12 months
  Minnesota Living with Heart Failure questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Wah David Siu, Professor, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Pokfulam, Hong Kong Island, Hong Kong

IPD SHARING:
Plan to Share IPD: No